CLINICAL TRIAL: NCT05889624
Title: Cognitive Behavioral Therapy Via Telehealth + Amitriptyline Compared to Cognitive Behavioral Therapy Via Telehealth: Pediatric Migraine Prevention (Responding With Evidence and Access for Childhood Headaches)
Brief Title: Responding With Evidence and Access for Childhood Headaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REACH Study; MP-2021C3-24936 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-05-10; First posted 2023-06-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Headache; Headache Disorders; Headache, Migraine; Migraine; Migraine Disorders; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: headache; migraine; cognitive behavioral therapy; pediatrics; diaphragmatic breathing; progressive muscle relaxation; imagery; relaxation; biofeedback
MeSH Terms: conditions — Headache; Headache Disorders; Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Cognitive Behavioral Therapy; Amitriptyline

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the principal investigator will remain blinded to the randomization assignment. All other study staff including the project manager, assistant project manager, study statistician, site investigators and study staff, participants, and their parents will be aware of the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT while taking a clinically-prescribed, pill-based prevention therapy (amitriptyline) (Experimental): This intervention consists of Cognitive Behavioral (CBT), a mind and body based intervention using education on gate control theory of pain, behavioral strategies such as muscle relaxation, activity pacing, and cognitive strategies including distraction, problem solving, and using calming self-statements. This arm will also take a daily oral dose of Amitriptyline, which will be clinically prescribed and managed by the patient's headache provider.
  Interventions: Behavioral: CBT; Drug: Amitriptyline
- CBT alone (Experimental): This intervention arm consists of 6 Cognitive Behavioral Therapy (CBT), a mind and body based intervention using education on gate control theory of pain, behavioral strategies such as muscle relaxation, activity pacing, and cognitive strategies including distraction, problem solving, and using calming self-statements.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — During an 8-week active treatment, participants will receive 6 telehealth CBT sessions, followed by a maintenance phase (16 weeks) when participants will receive 3 "booster" CBT sessions. The sessions will be conducted by teletherapists from the Clinical Coordinating Center at Cincinnati Children's using a standardized treatment manual. A parent/legal guardian will be included in 2 sessions teaching ways to be active coaches, encouraging use of effective coping skills and refraining from reinforcement of maladaptive coping. Each session will be about 45 minutes.
  Other Names: Cognitive Behavioral Therapy
Drug: Amitriptyline — During an 8-week active treatment, participants will begin taking a daily pill (amitriptyline) prescribed and managed clinically by the site headache provider. Amitriptyline will be taken once a day before bedtime. The weight based dosage will gradually be increased based on tolerability and a standardized titration protocol during the 8 week active treatment. The participant will remain on a maximum tolerated dose for the final 16 weeks (maintenance).
  Arms: CBT while taking a clinically-prescribed, pill-based prevention therapy (amitriptyline)

SUMMARY:
This comparative effectiveness study will clarify current first-line preventive treatment approaches for use by neurologists, psychologists, and primary care providers in the context of real world care, and will demonstrate the feasibility of Cognitive Behavioral Therapy (CBT) via telehealth for youth with migraine. The focus is on applying evidence-based care and enhancing access to it. CBT via telehealth while taking a clinically-prescribed, pill-based prevention therapy (amitriptyline) will be compared to CBT via telehealth alone.

DETAILED DESCRIPTION:
Migraine is the second most disabling disease in the world. Research has primarily focused on treating migraine in adults; however, approximately 10% of children and adolescents have migraine, suggesting that up to 7 million youth are impacted in the United States alone. Given that the majority of youth have migraine symptoms that persist into adulthood, there is a critical need to identify and improve access to the most effective preventive migraine treatments for this population as a means of reducing the long-term healthcare burden and functional impairment of this illness.

This comparative effectiveness study will test CBT while taking a clinically-prescribed, pill-based prevention therapy (amitriptyline) to CBT alone.

Participants will be involved in the study for approximately 28 weeks, with the first 4 weeks being a baseline period and the next 8 weeks involving six telehealth CBT sessions for both study groups (CBT while taking a clinically-prescribed pill-based prevention therapy [amitriptyline] compared to CBT alone), and dose titration of clinically-prescribed medication (amitriptyline) for the CBT + clinically-prescribed, pill-based prevention therapy (amitriptyline) group. During the remaining 16 weeks the participants will maintain the dose of medication (in the CBT + clinically-prescribed, pill-based prevention therapy (amitriptyline) group) and attend "booster" CBT sessions held three times over 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Migraine with or without aura that meets the International Classification of Headache Disorders (ICHD) criteria 5 or presentation of continuous headache that includes migranous episodes based upon headache history obtained by site PI or designee. (includes presentation with or without medication overuse headache as well)
* Headache Frequency: 4 or more headache days based upon prospective headache diary of 28 days prior to randomization
* Amitriptyline Eligible: Site PI or medical staff determined participant to be eligible for clinical prescription of amitriptyline as a preventive treatment for migraine
* English fluency: Able to complete the study visits and questionnaires in English

Exclusion Criteria:

* Current treatment includes amitriptyline and/or CBT specific to headache care
* Current prescribed preventive antimigraine medication within a period equivalent to < 5 half-lives of that medication before entering the baseline phase
* Current treatment with onabotulinumtoxinA (Botox) or CGRP-based monoclonal antibody medications for migraine prevention
* Youth who are pregnant
* Report of current or ongoing suicidal thoughts. Suicide attempt within the past six months. History of bipolar disorder, prolonged QT, or pre-existing significant constipation or gastroparesis
* Any and all other diagnoses or conditions which, in the opinion of the site investigator, would prevent the patient from being a suitable candidate for the study or interfere with the medical care needs of the participant

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in number of headache days | baseline to weeks 4-8 to weeks 20-24 (post treatment)
  This outcome measures whether there is a 50% reduction in the number of headaches days based on a self reported daily headache diary, per 28-day period, between the two arms.
Reduction to a PedMIDAS score of 20 or less | baseline to weeks 20-24 (post treatment)
  The PedMIDAS scale which evaluates the impact of headaches in school, home, play, and social activities, is comprised of six items that pertain to days missed in various activities over the past 90 days. Questions are answered by the youth in consultation with their parents and reviewed by study staff. The PedMIDAS scale is administered at baseline (covering the three months prior to enrollment) and at the endpoint visit (covering last three months of enrollment).
  This outcome measures whether there is a reduction in migraine related disability measured by the Pediatric Migraine Disability Scale (PedMIDAS) between the two arms. A reduction to a score of 20 or less, indicating mild impact of less is a meaningful outcome for patients and families and considered clinically significant.

SECONDARY OUTCOMES:
Change in absolute headache disability score on PedMIDAS | baseline to weeks 20-24 (post treatment)
  The PedMIDAS scale which evaluates the impact of headaches in school, home, play, and social activities, is comprised of six items that pertain to days missed in various activities over the past 90 days. Questions are answered by the youth in consultation with their parents and reviewed by study staff. The PedMIDAS scale is administered at baseline (covering the three months prior to enrollment) and at the post treatment visit (covering last three months of enrollment).
  A total PedMIDAS score (sum of items 1-6) was used in this study. Scores range from 0-240; with a score of 0-10 indicating no disability, 11-30 mild disability, 31-50 moderate disability, and more than 50 severe disability in daily activities.
Change in absolute headache days | baseline to weeks 4-8 to weeks 20-24 (post treatment)
  This outcome measures whether there is an absolute reduction in the number of headaches days based on a self reported daily headache diary, per 28-day period, between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Powers, PhD, Principal Investigator — Cincinnati Childrens Medical Center, Cincinnati
Locations (14):
- United States (14):
  - University of Alabama at Birmingham Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Colorado/Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Health System, Wilmington, Delaware
  - Clinical Integrative Research Center of Atlanta, Inc, Atlanta, Georgia
  - University of Louisville Health/Norton, Louisville, Kentucky
  - Louisiana State Univ/Children's Hospital of New Orleans, New Orleans, Louisiana
  - Dent Neurological Institute, Amherst, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Childrens, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center/ LeBonheur Children's Hospital, Memphis, Tennessee
  - Marshall Health, Huntington, West Virginia